CLINICAL TRIAL: NCT06218277
Title: Rapid Antimicrobial Susceptibility Testing with MIC Directly from Positive Blood Cultures with ASTar
Acronym: RASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2022-0379
Record Dates: First submitted 2023-12-18; First posted 2024-01-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bacteremia
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Intervention Model Description: Prospective in one group of patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ASTAR (Experimental): Use of the early AST results for guidance of the antimicrobial therapy
  Interventions: Diagnostic Test: ASTAR

INTERVENTIONS:
Diagnostic Test: ASTAR — Rapid AST with ASTAR

SUMMARY:
The investigators want to investigate the clinical impact of early antimicrobial susceptibility results for gram negative bacilli isolated from blood cultures on antimicrobial choices and early switches of antimicrobial therapy.

DETAILED DESCRIPTION:
Sepsis and septic shock are defined as a (life-threatening) organ dysfunction caused by an (uncontrolled) host response to an infection. Sepsis remains a leading cause of morbidity and mortality worldwide. In addition, sepsis is also associated with prolonged hospitalization and additional healthcare costs.

Sepsis and septic shock can be caused by a bloodstream infection. If bloodstream infection is suspected, blood cultures are collected.

In recent years, various devices and methods have been developed to make an antibiogram possible after a few hours, instead of the next day. The Q-linea AStar system will be used for this purpose in the medical microbiology laboratory. In contrast to the classic method, blood from the blood culture is not grafted onto a growth medium, but this blood is placed in a specific cartridge on the device, after which automatic sample processing takes place, which after six hours leads to a definitive susceptibility result for a large number of gram-negative bacilli and causes of bloodstream infections. Moreover, the reported antibiogram is not based on disk diffusion but on 'broth' microdilution (ISO 2776-1) where the sensitivity to a specific antibiotic is determined on the basis of a dilution series. This method allows sensitivity to be reported not only qualitatively (sensitive or resistant), but also allows reporting of the minimum inhibitory concentration (MIC value). This is the lowest concentration of an antibiotic at which the growth of the bacteria is inhibited and this fact allows the dose administered to be optimized if necessary.

The aim of this study is therefore, if this new method can be implemented, to retrospectively determine whether making the antibiogram more quickly available in the epidemiological setting of Ghent University Hospital offers added value: does the early available information lead to necessary and beneficial antibiotherapy changes or does the traditional diagnosis with reporting one day later prove to be equivalent? If the new working method were to lead to a clinically significant improvement in the established policy, this could necessitate an organizational adjustment in the operation of the laboratory.

To gain insight into this, clinical data will be collected during the study period necessary to evaluate the extent to which the faster results have had an impact on the antibiotherapy. There is therefore no need for additional sample collection from the patient. All collected data result from the standard hemoculture taken due to fever and/or frissons and concern clinical data that is routinely collected to formulate antibiotic recommendations for patients with positive hemocultures.

The following data will be collected pseudonymised for samples processed according to the new best practice:

* sample number
* gender and year of birth, date of sample inclusion
* presumed source of infection, empirically administered antibiotic
* time-to-positivity of the blood culture bottle (TTP), type blood culture bottle
* result of gram stain & duration until reporting, any antibiotic change based on. gram stain
* causative germ and resistance profile (e.g. ESBL, Multi-Drug Resistant P.aeruginosa, ...)
* result of antibiogram & duration until reporting (both methods), formulated advice, any antibiotic change based on. initially formulated advice (effect on antibiotic decision making), if necessary, additional advice and their associated impact on antibiotic policy
* time-to-first effective antibiotherapy, time-to-effective antibiotherapy based on antibiogram, time-to-optimal antibiotherapy, time-to-stop antibiotherapy, number of antibiotic days, antibiotic exposure (different classes for example), duration of empirical treatment (with T0 collection time of the hemoculture)

ELIGIBILITY:
Inclusion Criteria:

Patients with blood culture positive with gram negative bacilli

-

Exclusion Criteria:

* Mixed blood culture positivity on Gram stain
* Positive blood culture with gram negative bacilli in the previous 7 days
* Life expectancy of < 48 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Time tot first effective antibiotic therapy | 24 hours
  Time tot first effective antibiotic therapy

SECONDARY OUTCOMES:
Time to optimal antibiotic therapy | 72 hours
  Time to optimal antibiotic therapy
Number of different antibiotic classes used in treatment | 14 days
  Number of different antibiotic classes used in treatment
Time to stop antibiotic therapy | 14 days
  Time to stop antibiotic therapy
Time of empiric treatment | 72 hours
  Time of empiric treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jerina Boelens, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Messiaen AS, Vandendriessche S, De Muynck E, Strubbe G, De Bus L, Schelstraete P, Decommer K, De Smet S, Soetens A, Naesens L, Timmermans K, De Waele JJ, Veld DHI', Boelens J. Impact of reporting rapid susceptibility results in Gram negative bloodstream infections: a real world prospective study. Eur J Clin Microbiol Infect Dis. 2025 Apr;44(4):847-853. doi: 10.1007/s10096-025-05046-3. Epub 2025 Jan 25. PMID 39862301